CLINICAL TRIAL: NCT00037388
Title: Pediatrics:Chlamydia, Sickle Cell Anemia and Stroke Risk - Ancillary to STOP II
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1167; R01HL069114 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2008-01

CONDITIONS: Blood Disease; Anemia, Sickle Cell; Chlamydia Infections; Cerebrovascular Accident
MeSH Terms: conditions — Hematologic Diseases; Anemia, Sickle Cell; Chlamydia Infections; Stroke

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
To establish a link among Chlamydia infection, sickle cell anemia, and stroke risk.

DETAILED DESCRIPTION:
BACKGROUND:

Infection with Chlamydia pneumoniae (C. pneumoniae) is associated with an increased risk of cerebrovascular disease in the general population. Children with sickle cell anemia (SCA) are 200 times more likely to have cerebrovascular disease than normal children and are known to have an altered immune response to many infectious pathogens. C. pneumoniae is the leading infectious cause of acute chest syndrome which, interestingly, is a well- established risk factor for stroke in children with SCA. Preliminary data indicates that SCA patients with magnetic resonance imaging (MRI)-documented cerebral infarction are 12 times more likely to have C. pneumoniae infection than SCA patients with normal MRI scans. The investigators hypothesize that SCA patients have an abnormal immune response to C. pneumoniae that results in persistent infection which, in turn, triggers the development of cerebrovascular disease. Sickle cell anemia patients with an elevated velocity on transcranial doppler ultrasound (TCD) are known to be at high risk to develop stroke and an elevated TCD likely reflects underlying vascular disease. In addition, the Stroke Prevention in Sickle Cell Anemia Trial (STOP) demonstrated that almost 40 percent of children with an elevated TCD have evidence of cerebral infarction on MRI. Children with abnormal TCDs are, therefore, an appropriate population to investigate an association between cerebrovascular disease and C. pneumoniae infection.

The study is in response to an initiative on Ancillary Studies in Heart, Lung, and Blood Disease Trials released in June, 2000.

DESIGN NARRATIVE:

The study is ancillary to the STOP II clinical trial. The intent is: 1) To determine if C. pneumoniae infection is associated with cerebral infarction in children with SCA; 2) To characterize the immunological response to C. pneumoniae infection in patients with SCA. Establishing a link between C.pneumoniae infection and cerebral infarction will open the door to novel, less toxic approaches to the treatment and prevention of stroke in SCA, including antibiotics and vaccines.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2004-07; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Styles — UCSF Benioff Children's Hospital Oakland